CLINICAL TRIAL: NCT00196092
Title: Zenith® AAA Endovascular Graft Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99-514
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2007-12

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Surgical Procedures, Operative; Compassionate Use Trials; Therapeutics

ARMS (8):
- 1 (Other): Roll-in
  Interventions: Device: Roll-in
- 2 (Other): Surgical
  Interventions: Device: Surgical
- 3 (Other): Standard Risk
  Interventions: Device: Standard Risk
- 4 (Other): High Risk
  Interventions: Device: High Risk
- 5 (Other): Compassionate Use
  Interventions: Device: Compassionate Use
- 6 (Other): Treatment for females.
  Interventions: Device: Treatment for females
- 7 (Other): Standard Risk Continued Access
  Interventions: Device: Standard Risk Continued Access
- 8 (Other): High Risk Continued Access
  Interventions: Device: High Risk Continued Access

INTERVENTIONS:
Device: Roll-in — Proctored entry.
  Arms: 1
Device: Surgical — Surgery
  Arms: 2
Device: Standard Risk — Standard Endovascular repair
  Arms: 3
Device: High Risk — High Risk Endovascular repair.
  Arms: 4
Device: Compassionate Use — Endovascular repair for compassionate use patients.
  Arms: 5
Device: Treatment for females — Endovascular repair in female patients
  Arms: 6
Device: Standard Risk Continued Access — Continued Access Endovascular repair for standard risk patients.
  Arms: 7
Device: High Risk Continued Access — Continued Access Endovascular Repair for High Risk Patients.
  Arms: 8

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Cook Zenith Endovascular Graft for the treatment of abdominal aortic (AAA), aortoiliac, and iliac aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an aortic or aortoiliac aneurysm with diameter greater than or equal to 4 cm.
2. Patients with an iliac aneurysm with diameter greater than or equal to 3.5 cm.
3. Patients with an aortic, aortoiliac, or iliac aneurysm with a history of growth greater than or equal to 0.5 cm per year.

Exclusion Criteria:

1. Patients less than 18 years of age.
2. Patient with a life expectancy less than 2 years.
3. Patients who are pregnant.
4. Patients unwilling to comply with the follow-up schedule.
5. Patient inability or refusal to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 819 (Actual)
Dates: Start 2000-01; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Greenberg, M.D., Principal Investigator — The Cleveland Clinic